CLINICAL TRIAL: NCT04036864
Title: Retrospective Study of Singing-voice Disorders and Aerodynamic Profiles in Dysodic Singers
Brief Title: Singing-voice Disorders and Aerodynamic Profiles in Dysodic Singers
Acronym: AeroDysodiaPro
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: GIPSA-lab, Grenoble, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0339
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Dysodia
Keywords: Singers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Singers are over-represented in phoniatric consultation; they present increased risk of developing voice disorders. They represent a specific population among phoniatric patients (specific singing-voice complaints, increased sensitivity to voice). Singing-voice disorder is called dysodia in the same way as dysphonia, which refers to speaking-voice disorders. The diagnosis of dysodia is made after a laryngeal examination and a voice assessment to identify patient's speech and singing difficulties. Most studies on prevalence of voice disorders in singers come from the American continent. Very few descriptions of this population have been made in France.

Voice assessment of dysodic singers includes aerodynamic voice measurements. The use of aerodynamic measurements for the diagnosis of voice pathologies is now widely demonstrated. These parameters include measurements of estimated subglottal pressure (ESGP), phonation threshold pressure (PTP) (minimum pressure to initiate a sound) and oral airflow (OAF). They depend on the level of training of singers and the type of vocal dysfunction. Aerodynamic behaviours of dysodic singers have not yet been described, although they can help to better identify the singer's vocal difficulties and could be essential parameters for targeting more precisely rehabilitation exercises proposed in voice therapy.

This study aims to describe the characteristics of a French population of singers consulting in phoniatrics and their aerodynamic behaviours. Do the singers' aerodynamic parameters (pressure, flow) reflect the dysfunctions in singing voice? Based on results of the literature on speaking and singing non-pathological voice, the investigators hypothesize that during voice assessment, ESGP values will be increased and OAF ones will be decreased over the entire vocal range of the singer in case of voice pathology.

DETAILED DESCRIPTION:
Singers are over-represented in phoniatric consultation; they present increased risk of developing voice disorders whether they are amateurs or professionals. They represent a specific population among phoniatric patients because of their increased sensitivity to the slightest voice change that makes them consult earlier than non-. In addition, their complaints are specific to singing voice. The most common lesion found in singers is vocal-fold nodule. It comes from a vocal straining characterized by the use of a pressed phonation mode, resulting in an increased subglottal pressure and a decreased flow rate.

Singing-voice disorder is called dysodia in the same way as dysphonia, which refers to speaking-voice disorders. Dysodia results in a variety of symptoms. Acoustic signs are the most numerous: tonal anomalies (lack of accuracy, reduction of vocal range); dynamic anomalies (problem to sing softly or loudly); timbre abnormalities (vibrato problems, strained voice, roughness, difficulties on attacks). Dysodia also results in respiratory disorders, physical signs, psychological consequences and damage to hedonistic properties (loss of comfort, vocal endurance, musicality). It can reach amateur or professional singers. For professional singers, voice is the main working tool. When they have dysodia, professional difficulties can be temporary or even lead to the loss of work. In addition, dysodia can lead to financial loss and well-documented anxiety. For amateur singers, dysodia hinders their musical practice, thus limiting the recognized benefits of choral singing on cohesion, social integration and personal development. The diagnosis of dysodia is made after a laryngeal examination and a vocal assessment to identify patient's speech difficulties.

Voice assessment includes subjective voice analyses but also instrumental analyses that include acoustic, electrophysiological and aerodynamic voice measurements. The interest of aerodynamic parameters for the diagnosis of vocal pathologies is now widely demonstrated. These parameters include measurements of estimated subglottal pressure (ESGP), phonation threshold pressure (PTP) (minimum pressure to initiate a sound) and oral air flow (OAF). They depend on the level of training of singers and the type of vocal dysfunction. These aerodynamic data are collected with devices such as the Assisted Voice Evaluation Device (EVA2©) used in the laryngeal department of the Gui de Chauliac University Hospital. These pressure and flow parameters are higher in opera singers than in non-singers. In clinical practice, the ESGP and PTP are higher during vocal straining in dysphonic patients. Concerning OAF, results remain controversial: increase with vocal effort in euphonics non-singers; decrease with intensity increase in euphonic non-singers. Aerodynamic behaviours of dysodic singers have not yet been described, although they can help to better identify the singer's vocal difficulties and could be essential parameters for targeting more precisely rehabilitation exercises proposed in voice therapy.

In addition, most studies on prevalence of vocal disorders in singers come from the American continent. Very few descriptions of this population have been made in France. The few that exist are quite old or involve limited samples. Moreover, to date, no study has explored the aerodynamic profiles (flow and pressure) of singers, although these profiles are considered to be relevant clinical indicators to describe the singer's vocal difficulties and thus precise more specific therapeutic objectives.

In this context, our project aims to fill these gaps by describing a French population of singers consulting in phoniatrics and describing their aerodynamic behaviours. Do the singers' aerodynamic parameters (pressure, flow) reflect the dysfunctions in singing voice? Based on results of the literature on speaking and singing non-pathological voice, the investigators hypothesize that during voice assessment, the values of ESGP and PTP will be increased and that those of OAF will be decreased over the entire range of the singer in case of vocal pathology

ELIGIBILITY:
Inclusion Criteria:

* have consulted Dr Amy de la Bretèque, phoniatrist, between January 2015 and June 2018
* be a singer (professional or amateur)
* be over 18 years old

Exclusion Criteria:

* under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have consulted the phoniatrician (Dr Amy de la Bretèque) of the ENT department of the Gui de Chauliac hospital between January 2015 and June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Aerodynamic data : estimated subglottal pressure | 1 day
  estimated subglottal pressure (values in hPa)
Aerodynamic data : phonation pressure threshold | 1 day
  phonation pressure threshold (values in hPa)
Aerodynamic data : oral airflow rate | 1 day
  oral airflow rate (values in l/s).

SECONDARY OUTCOMES:
social and medical data : age | 1 day
  age (yo)
social and medical data : sex | 1 day
  sex (male or female)
social and medical data : occupation | 1 day
  occupation : profession noted in the file by the phoniatrician
social and medical data : singing style | 1 day
  singing style : opera, concert/oratorio/recital, recording artist, pop, rock, jazz, gospel and soul, country and western, world music, vocal groups, French commercial singing.
social and medical data : level of training | 1 day
  level of training : superstars, international singers, national/big city singers, regional/touring, local community (including semiprofessionals), full-time students of singing and amateur.
social and medical data : voice complaint | 1 day
  voice complaint : vocal difficulties reported by the patient to the phoniatrician and noted in the medical files
social and medical data : phoniatric diagnosis | 1 day
  phoniatric diagnosis : diagnosis by the phoniatrician specifying whether there are laryngeal lesions
social and medical data : tobacco consumption | 1 day
  tobacco consumption (yes or no, volume)
social and medical data : voice treatment | 1 day
  voice treatment : treatment proposed by the phoniatrician (no treatment, surgery, voice therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Marion BEAUD, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC